CLINICAL TRIAL: NCT00482950
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate Safety and Efficacy of PHX1149T in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate Safety and Efficacy of PHX1149T in Subjects With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Phenomix (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHX1149-Prot202
Expanded Access: Available
Record Dates: First submitted 2007-06-04; First posted 2007-06-06 (Estimated); Last update posted 2009-06-08 (Estimated); Status verified 2009-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PHX1149T

SUMMARY:
This study is to test the efficacy and safety of PHX1149T in combination with metformin, a glitazone, or metformin and a glitazone in subjects with Type 2 diabetes for 12 weeks. After completing the 12 week double blind part of the study, subjects can enter an open label extension study

ELIGIBILITY:
Key Entry Criteria:

* Type 2 diabetes mellitus, diagnosed at least 4 months but not more than 12 years prior to screening.
* Male and non-pregnant, non-lactating (and not planning to become pregnant during the study) female subjects with a BMI of 25 to 48 kg/m2, inclusive. For India the BMI is 23 to 48 kg/m2, inclusive.
* Current treatment of Type 2 diabetes mellitus with a stable dose of metformin of 1500 mg or more (or the highest tolerated dose), or TZD (any labeled dose), or metformin + TZD at doses used in accordance with product labeling for at least 4 weeks (metformin) or 10 weeks (TZD) prior to screening (Visit 1).
* Fasting plasma glucose of 118 - 220 mg/dL (6.6 - 12.2 mmol/L), inclusive; HbA1c 7.3% - 11.0%, inclusive; and a fasting plasma C peptide greater than 0.26 nmol/L at screening. For Argentina the allowed upper limit of HbA1c is ≤ 10.5%. For Canada the upper limit will be 10.0%
* No Type 1 diabetes mellitus or marked diabetic long-term complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-04; Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Guler, MD, Study Director — Phenomix Corp.
Locations (26):
- United States (22):
  - Chula Vista, California
  - Fullerton, California
  - Long Beach, California
  - Orange, California
  - Kissimmee, Florida
  - Melbourne, Florida
  - Bloomington, Indiana
  - Wichita, Kansas
  - Kansas City, Missouri
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Trenton, New Jersey
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Medford, Oregon
  - Westminster, Pennsylvania
  - Columbia, South Carolina
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
- Multiple Cities, Argentina
- Mutiple Cities, Canada
- Mutiple Cities, India
- Mutiple Cities, Mexico